CLINICAL TRIAL: NCT06895512
Title: A Randomized, Double-blind, Parallel-controlled, Multicenter, Phase III Study to Evaluate the Efficacy and Safety of HLX15-IV Versus DARZALEX® in Combination with Lenalidomide-Dexamethasone (Rd) in Transplant-ineligible Patients with Newly Diagnosed Multiple Myeloma
Brief Title: A Study to Evaluate the Efficacy and Safety of HLX15-IV Versus DARZALEX® in Combination with Lenalidomide-Dexamethasone (Rd) in Transplant-ineligible Patients with Newly Diagnosed Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX15-IV-NDMM-301
Record Dates: First submitted 2025-03-10; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Newly Diagnosed Multiple Myeloma
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HLX15-IV-Rd (Experimental): HLX15-IV in combination with Lenalidomide-Dexamethasone (Rd)
  Interventions: Drug: HLX15-IV
- DARZALEX-Rd (Active Comparator): DARZALEX in combination with Lenalidomide-Dexamethasone (Rd)
  Interventions: Drug: Darzalex

INTERVENTIONS:
Drug: HLX15-IV — recombinant anti-CD38 human monoclonal antibody injection
  Arms: HLX15-IV-Rd
Drug: Darzalex — recombinant anti-CD38 human monoclonal antibody injection
  Arms: DARZALEX-Rd

SUMMARY:
This is a randomized, double-blind, parallel-controlled, multicenter, phase III study to compare the efficacy and safety of HLX15-IV in combination with Rd (HLX15-IV-Rd) versus DARZALEX® in combination with Rd (D-Rd) in patients with NDMM who are ineligible for autologous stem cell transplantation (ASCT).

ELIGIBILITY:
Inclusion Criteria:

1. Capable to understand and sign the ICF.
2. Patients aged ≥ 18 years .
3. Patient must have documented multiple myeloma (MM) satisfying the International Myeloma Working Group (IMWG) diagnostic criteria for MM.
4. Newly diagnosed, untreated and not considered candidate for autologous stem cell transplantation (ASCT).
5. Patient must have an ECOG performance status score of 0.
6. Patient must have pretreatment clinical laboratory values.
7. Contraceptive use by men or women should be consistent with local regulations.
8. A WOCBP must have a negative serum pregnancy test at screening within 72 hours prior to randomization.

Exclusion Criteria:

1. Patient has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), Waldenström's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
2. Patient has plasma cell leukemia or POEMS syndrome .
3. Patient has prior or current systemic therapy or ASCT for MM before randomization.
4. Patient has peripheral neuropathy or neuropathic pain Grade 2 or higher.
5. Patient has a history of malignancy (other than MM) within 3 years before randomization .
6. Patient has clinical signs of meningeal involvement of MM.
7. Patient has known COPD, persistent asthma, or a history of asthma within the last 2 years.
8. Patient is known to be seropositive for history of human immunodeficiency virus (HIV) or known to have treponema pallidum antibodies (Anti-TP).
9. Patient is known to have active hepatitis B or C.
10. Patient has any concurrent medical or psychiatric condition or disease that is likely to interfere with the study procedures or results.
11. Patient has clinically significant cardiac disease.
12. Patient has known allergies, hypersensitivity, or intolerance to treatment drugs.
13. Patient has history of drug abuse or substance abuse.
14. Patient is a woman who is pregnant, or breast-feeding, or planning to become pregnant or donate eggs (ova, oocytes).
15. Patient had radiation therapy within 14 days of randomization.
16. Patient had plasmapheresis within 28 days of randomization.
17. Patient had major surgery within 28 days before randomization.
18. Patient in clinical trials of any other drug or device within 3 months before randomization.
19. Patient has any condition could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
IRC-assessed Week 24 rate of very good partial response (VGPR) or better | 24 weeks
  the percentage of patients achieving VGPR or CR (including sCR) until Week 24 after the date of randomization.

SECONDARY OUTCOMES:
Investigator-assessed Week 24 rate of VGPR or better | 24 weeks
  the percentage of patients achieving VGPR or CR (including sCR) until Week 24 after the date of randomization
IRC- and investigator-assessed Week 12, 36 and 48 rate of VGPR or better | 12,36,48 weeks
  percentage of patients achieving VGPR or CR (including sCR) until Week 12, 36 and 48 after the date of randomization
IRC- and investigator-assessed partial response (PR) rate | 48 weeks
  the percentage of patients achieving PR at any time point after the date of randomization
IRC- and investigator-assessed complete response (CR) rate | 48 weeks
  the percentage of patients achieving CR at any time point after the date of randomization.
IRC- and investigator-assessed stringent complete response (sCR) rate | 48 weeks
  percentage of patients achieving sCR at any time point after the date of randomization
IRC- and investigator-assessed complete response (CR) or better rate | 48 weeks
  the percentage of patients achieving CR or sCR at any time point after the date of randomization.
IRC- and investigator-assessed overall response rate | 48 weeks
  the percentage of patients who achieve PR or better after the date of randomization.
IRC- and investigator-assessed time to response (TTR) | 48 weeks
  the time from the date of randomization to the date of initial documentation of a response (PR or better) for patient who had achieved a response of PR or better
IRC- and investigator-assessed duration of response (DOR) | 48 weeks
  the date of initial documentation of a response (PR or better) to either progressive disease according the IMWG criteria, or death, whichever occurs first
IRC- and investigator-assessed progression free survival (PFS) | 48 weeks
  the duration from the date of randomization to either progressive disease, according to the IMWG response criteria, or death, whichever occurs first.
Minimal residual disease (MRD) negative rate | 48 weeks
  the percentage of patients who achieve negative MRD at least once during the confirmed complete response (CR) or better according to the IMWG response criteria.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Health Status (EORTC-QLQ-C30). | 48 weeks
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Health Status (EORTC-QLQ-C30).Minimum and maximum values is according to the items, the score range of item 1-28 is 1-4, the score range of item 29-30 is 1-7. The higher the overall score is, the better the overall quality of life is.
EuroQoL 5-Dimension 5-Level Health Status (EQ-5D-5L) Questionnaire. | 48 weeks
  EuroQoL 5-Dimension 5-Level Health Status (EQ-5D-5L) Questionnaire.The description of health status is divided into five levels.Health Status Index range is -0.59-1.00, VAS range is 0-100.The higher the Health Status Index and VAS score are, the better the health condition is; the lower the dimension description score is, the fewer problems there are.
Incidence and severity of adverse events (AEs) | 52 weeks
  severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version [v] 5.0, vital signs and clinical laboratory test results
Time to reach maximum serum drug concentration at steady state (Tmax, ss) | 48 weeks
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Time to reach maximum serum drug concentration(Tmax) | 48 weeks
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Immunogenicity | 48 weeks
  Incidence of ADA and/or NAb for HLX15-IV and DARZALEX

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hospital, Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No